CLINICAL TRIAL: NCT02056522
Title: Non-invasive Melanoma Assessment Using a Topical Fluorescence Reagent and Optical Imaging: the MDS (Melanoma Detecting System)
Brief Title: Non-invasive Melanoma Assessment Using a Topical Fluorescence Reagent and Optical Imaging
Status: Completed | Type: Observational
Sponsor: Orlucent, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: OMS 001
Record Dates: First submitted 2013-12-15; First posted 2014-02-06 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2018-02

CONDITIONS: Skin Lesions
Keywords: Melanoma; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Suspicious skin lesions.: No intervention is administered.

SUMMARY:
The use of MDS to access the presence of melanoma in the skin.

DETAILED DESCRIPTION:
A topical agent is applied to suspicious skin lesions and imaged. The images are analyzed to provide a score that correlates with the probability for the presence of melanoma in the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with skin lesion with one or more of the ABCDE features and recommended for a skin biopsy.
* The lesion is accessible to the imaging device, with at least 1 cm of skin around the lesion that is accessible to the MDS.
* Male and female ≥ 21 years old.
* Subject is capable of giving written informed consent.
* Primary excision.

Exclusion Criteria:

* The lesion is less than 1 cm from the eyes.
* The lesion is on the palms of hands or soles of the feet.
* Mucosal lesion.
* Pregnant females.
* Low study procedure compliance.
* Patients who are mentally or physically unable to comply with all aspects of the study.
* Undergoing chemotherapy.
* Minor or legally incompetent and not able to sign the consent form.
* Patient previously tested by MDS and was diagnosed with melanoma during the study.

Ages: 21 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individual referred by a dermatologist or plastic surgeon for a skin biopsy or lesion excision.
Sampling Method: Probability Sample
Enrollment: 357 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
To validate the performance of MDS | 28 days

SECONDARY OUTCOMES:
To calculate and specify the PPV and NPV of the MDS for melanoma detection when used as an adjacent tool to visual skin examination. | 28 days

OTHER OUTCOMES:
To further establish the safety of the MDS. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Shokrey Kassis, MA, Principal Investigator — Head of Plastic Surgery
Locations (2):
- Israel (2):
  - Clalit Health Services, Kiryat Bialik
  - Ziv Medical Center, Safed

IPD SHARING:
Plan to Share IPD: Undecided